CLINICAL TRIAL: NCT00149240
Title: A Phase II, Multicentre, Randomised, Double-blind, Parallel and Controlled With Placebo Pilot Study to Evaluate the Efficacy and Safety of a Single Dose of Botulinum Toxin Type A (Dysport) Associated With Rehabilitation Treatment, in Patients With Primary Myofascial Syndrome of Cervical and Dorsal Localisation
Brief Title: Botulinum Toxin Type A (Dysport) Associated With Rehabilitation Treatment in Patients With Primary Myofascial Pain Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-92-52120-089; 2004-001443-29 (EudraCT Number)
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Myofascial Pain Syndromes
Keywords: DYSPORT; botulinum toxin A; myofascial pain syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Biological: Botulinum toxin type A

SUMMARY:
The main purpose of this study is to determine the effectiveness and safety of one dose of botulinum toxin type A (Dysport) associated with rehabilitation treatment on pain control in patients with a type of back pain called primary myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary myofascial pain syndrome of cervical and dorsal localization, less than two years of length, who must have been diagnosed with the evidence of "trigger points" in which conventional treatment with oral analgesia, rehabilitation and local anesthesia has not been clinically successful for more than 15 days.
* Punctuation of 4cm or more in a 10cm visual analog scale.
* Previous positive response (self-limited reduction -less than 15 days- of pain) after an anaesthetic infiltration in the trigger point.

Exclusion Criteria:

* Patients diagnosed with fibromyalgia or with a spread pain.
* Patients having received previously botulinum toxin.
* Patients having received anesthetic injections at the trigger points within the month before the visit.
* Patients having received corticosteroids injections at the trigger points within three months before the selection visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01; Primary Completion 2006-02-02 (Actual); Study Completion 2006-02-02 (Actual)

PRIMARY OUTCOMES:
The following parameters are measured at Inclusion, Week 2, Week 4, Week 8 and Week 12 of the study:
Pain evaluated by the Investigator through the determination of threshold of pain by pressure algometry for each trigger point.
Pain evaluated by the patient through a visual analog scale.
Evaluation of the Clinical Global Impressions of Change by the Investigator and by the patient.
Usual analgesic intake modification (on a daily basis by filling out a Patient's diary).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (4):
- Spain (4):
  - University Hospital "Vall d 'Hebrón". Barcelona, Barcelona
  - University Hospital of Alcorcón, Madrid
  - Complexo Médico Quirúrgico del Conxo, Santiago de Compostela
  - University Hospital "La Fe". Valencia, Valencia